CLINICAL TRIAL: NCT07193849
Title: Impact of Using Zinc Oxide Versus Moist Exposed Wound Ointment (MEBO) in Treatment of Second Stage Pressure Ulcer: A Randomized Control Clinical Trial
Brief Title: Zinc Oxide VS MEBO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdullah Medical City (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1032; 23071104 (Other: Saudi Food and Drug Authority (SFDA))
Record Dates: First submitted 2025-06-29; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pressure Injury; Pressure Injury Stage 2; Bedsore; Pressure Ulcers Stage II; Pressure Ulcer, Buttock
Keywords: pressure injury; pressure ulcer; MEBO; Zinc oixid
MeSH Terms: conditions — Pressure Ulcer | interventions — Zinc Oxide

STUDY DESIGN:
Intervention Model Description: A randomized control clinical trial
Masking Description: no masking in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The zinc oxide group (Active Comparator): The zinc oxide group will receive topical zinc oxide twice every 12 hours daily
  Interventions: Drug: zinc oxide
- MEBO group (Active Comparator): patients in the MEBO group will receive topical MEBO ointment twice every 12 daily
  Interventions: Drug: MEBO Wound Ointment

INTERVENTIONS:
Drug: MEBO Wound Ointment — both are used for second pressure ulcer
  Arms: MEBO group
Drug: zinc oxide — both are used to treat second degree pressure ulcer but with no superiority
  Arms: The zinc oxide group

SUMMARY:
randomize control trial to evaluate the efficacy of using zinc oxide versus moist exposed wound ointment in treatment of second stage pressure ulcer.

DETAILED DESCRIPTION:
In this study the subject will be randomized using electronic randomization 1:1 ratio. The randomization list was generated electronically through R using the Random Allocation Rule. The data will be collected using Assessment sheet of patient with second stage pressure ulcer tool. Patients will equally be allocated into 2 groups randomly. The zinc oxide group will receive topical zinc oxide twice every 12 hours daily and patients in the MEBO group will receive topical MEBO ointment twice every 12 daily. Patient will be examined daily till complete healing for the pressure ulcer and maximum one month. The Bates-Jensen Wound Assessment Tool (BWAT) will be used to evaluate wound healing. It is a validated wound assessment tool which is used in many healthcare settings for wound assessment

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate.
* KAMC cases in medical ward, neuroscience ward, and intensive care unit.
* Newly cases diagnosed with second stage pressure ulcer according to the European pressure ulcer advisory panel/national pressure ulcer advisory panel (NPUAP) guidelines.

Exclusion Criteria:

* Not consenting to participate
* Patients with suspected hypersensitivity reactions to any of the topical formulation's ingredients.
* Either a category III or IV pressure ulcer.
* Evidence of deep tissue injury (exudative drainage, purple or maroon localized area of discolored intact skin or blood-filled blister due to pressure damage).
* Signs of wound infection (pus draining from the ulcer, a foul-smelling odour, tenderness, heat and increased redness in the surrounding skin and fever).
* Patients who undertaking other therapies that could affect healing, such as corticosteroids, radiation therapy, or chemotherapy for cancer.
* Heavy smoking (more than 20 cigarettes a day).
* Concomitant chronic disease (e.g., diabetes mellitus or frank vascular disease such as Buerger's disease).
* Patients who unable to continue the study because of death, discharge, or change in the care setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing | 30 days
  Wound healing will be assessed by using Bates-Jensen Wound Assessment Tool (BWAT) daily for both treatments.
  (BWAT) consists of 13 items to evaluate wound size, type and depth, Each item is graded on a scale of 1 to 5, where a score of 1 indicates progress toward healing while a score of 5 indicates the absence of healing or wound deterioration. Cumulative BWAT scores vary from 13 to 65

SECONDARY OUTCOMES:
Recovery time | 30 days
  The duration of treatment will be record at the assessment sheet so Recovery time will be determined from this sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ebtisam AbdElatif Ebrahim, Master degree of science in nu, Principal Investigator — King Abdullah Medical City in Holy Capital
Locations (1):
- King Abdulla Medical City in Holy capital, Mecca, Western Reagan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
we are still conducting the study after publication we might be interested and ready for sharing the full plan

REFERENCES:
- [Background] Andrade CC, Almeida CF, Pereira WE, Alemao MM, Brandao CM, Borges EL. Costs of topical treatment of pressure ulcer patients. Rev Esc Enferm USP. 2016 Apr;50(2):295-301. doi: 10.1590/S0080-623420160000200016. English, Portuguese. PMID 27384210
- [Background] Boyko TV, Longaker MT, Yang GP. Review of the Current Management of Pressure Ulcers. Adv Wound Care (New Rochelle). 2018 Feb 1;7(2):57-67. doi: 10.1089/wound.2016.0697. PMID 29392094
- [Background] Demarre L, Van Lancker A, Van Hecke A, Verhaeghe S, Grypdonck M, Lemey J, Annemans L, Beeckman D. The cost of prevention and treatment of pressure ulcers: A systematic review. Int J Nurs Stud. 2015 Nov;52(11):1754-74. doi: 10.1016/j.ijnurstu.2015.06.006. Epub 2015 Jun 25. PMID 26231383
- [Background] Qaseem A, Mir TP, Starkey M, Denberg TD; Clinical Guidelines Committee of the American College of Physicians. Risk assessment and prevention of pressure ulcers: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2015 Mar 3;162(5):359-69. doi: 10.7326/M14-1567. PMID 25732278
- [Background] Westby MJ, Dumville JC, Soares MO, Stubbs N, Norman G. Dressings and topical agents for treating pressure ulcers. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD011947. doi: 10.1002/14651858.CD011947.pub2. PMID 28639707
- [Background] VanGilder C, Amlung S, Harrison P, Meyer S. Results of the 2008-2009 International Pressure Ulcer Prevalence Survey and a 3-year, acute care, unit-specific analysis. Ostomy Wound Manage. 2009 Nov 1;55(11):39-45. PMID 19934462
- [Background] Gibbons W, Shanks HT, Kleinhelter P, Jones P. Eliminating facility-acquired pressure ulcers at Ascension Health. Jt Comm J Qual Patient Saf. 2006 Sep;32(9):488-96. doi: 10.1016/s1553-7250(06)32064-8. PMID 17987872
- [Background] Zaratkiewicz S, Whitney JD, Lowe JR, Taylor S, O'Donnell F, Minton-Foltz P. Development and implementation of a hospital-acquired pressure ulcer incidence tracking system and algorithm. J Healthc Qual. 2010 Nov-Dec;32(6):44-51. doi: 10.1111/j.1945-1474.2010.00076.x. PMID 20946425
- [Background] Li W, Ma Y, Yang Q, Pan Y, Meng Q. Moist exposed burn ointment for treating pressure ulcers: A multicenter randomized controlled trial. Medicine (Baltimore). 2017 Jul;96(29):e7582. doi: 10.1097/MD.0000000000007582. PMID 28723796
- [Background] Harris C, Bates-Jensen B, Parslow N, Raizman R, Singh M, Ketchen R. Bates-Jensen wound assessment tool: pictorial guide validation project. J Wound Ostomy Continence Nurs. 2010 May-Jun;37(3):253-9. doi: 10.1097/WON.0b013e3181d73aab. PMID 20386331
- [Background] Golden MH, Golden BE, Jackson AA. Skin breakdown in kwashiorkor responds to zinc. Lancet. 1980 Jun 7;1(8180):1256. doi: 10.1016/s0140-6736(80)91722-5. No abstract available. PMID 6104076
- [Background] Haley JV. Zinc sulfate and wound healing. J Surg Res. 1979 Sep;27(3):168-74. doi: 10.1016/0022-4804(79)90127-6. No abstract available. PMID 470359
- [Background] Jurjus A, Atiyeh BS, Abdallah IM, Jurjus RA, Hayek SN, Jaoude MA, Gerges A, Tohme RA. Pharmacological modulation of wound healing in experimental burns. Burns. 2007 Nov;33(7):892-907. doi: 10.1016/j.burns.2006.10.406. Epub 2007 May 22. PMID 17521821
- [Background] Wang QS, Tang QL, Zhang L, et al. MEBO for treating 47 cases of chronic ischemic ulcer in lower limber. Chin J Burns Wound Surface Ulcer 2005; 17:296-7. (In Chinese)
- [Background] National Pressure Ulcer Advisory Panel (NPUAP). PUSH Tool. Washington, DC: National Pressure Ulcer Advisory Panel; 2010
- [Background] Jewo PI, Fadeyibi IO, Babalola OS, Saalu LC, Benebo AS, Izegbu MC, Ashiru OA. A Comparative Study of the Wound Healing Properties of Moist Exposed Burn Ointment (MEBO) and Silver Sulphadiazine. Ann Burns Fire Disasters. 2009 Jun 30;22(2):79-82. PMID 21991159
- [Background] Li JH, Zhang L, Tang QL, et al. Clinical observation on effect of MEBO on neurogenic ulcer. Liaoning J Tradit Chin Med 2012; 39:1095-6. (In Chinese)
- [Background] Hirsch T, Ashkar W, Schumacher O, Steinstraesser L, Ingianni G, Cedidi CC. Moist Exposed Burn Ointment (MEBO) in partial thickness burns - a randomized, comparative open mono-center study on the efficacy of dermaheal (MEBO) ointment on thermal 2nd degree burns compared to conventional therapy. Eur J Med Res. 2008 Nov 24;13(11):505-10. PMID 19073386
- [Background] Yue J, Zhang Q, Sun Z, Du W, Yu C. A case of electroacupuncture therapy for pressure ulcer. Acupunct Med. 2013 Dec;31(4):450-1. doi: 10.1136/acupmed-2013-010418. Epub 2013 Aug 5. No abstract available. PMID 23917394
- [Background] Zhang QH, Yue JH, Li CR, Sun ZR. Moxibustion for the treatment of pressure ulcers: study protocol for a pilot, multicentre, randomised controlled trial. BMJ Open. 2014 Dec 30;4(12):e006423. doi: 10.1136/bmjopen-2014-006423. PMID 25550296
- [Background] Zhang QH, Yue JH, Sun ZR. Electroacupuncture for pressure ulcer: a study protocol for a randomized controlled pilot trial. Trials. 2014 Jan 6;15:7. doi: 10.1186/1745-6215-15-7. PMID 24393344
- [Background] Bhattacharya S, Mishra RK. Pressure ulcers: Current understanding and newer modalities of treatment. Indian J Plast Surg. 2015 Jan-Apr;48(1):4-16. doi: 10.4103/0970-0358.155260. PMID 25991879
- [Background] Yap TL, Kennerly SM, Horn SD, Bergstrom N, Datta S, Colon-Emeric C. TEAM-UP for quality: a cluster randomized controlled trial protocol focused on preventing pressure ulcers through repositioning frequency and precipitating factors. BMC Geriatr. 2018 Feb 20;18(1):54. doi: 10.1186/s12877-018-0744-0. PMID 29463211
- [Background] Coleman S, Smith IL, McGinnis E, Keen J, Muir D, Wilson L, Stubbs N, Dealey C, Brown S, Nelson EA, Nixon J. Clinical evaluation of a new pressure ulcer risk assessment instrument, the Pressure Ulcer Risk Primary or Secondary Evaluation Tool (PURPOSE T). J Adv Nurs. 2018 Feb;74(2):407-424. doi: 10.1111/jan.13444. Epub 2017 Sep 28. PMID 28833356
- [Background] Saghalein S, Dehghan K, Shadvar K, Mahmoodpoor A, Sanaie S, Ostadi Z. Bedsore: Epidemiology; Risk Factors; Classification; Assessment Scales and Management. Archives of Anesthesiology and Critical Care. 2016;2(3):226-30
- [Background] de Almeida Medeiros AB, da Conceicao Dias Fernandes MI, de Sa Tinoco JD, Cossi MS, de Oliveira Lopes MV, de Carvalho Lira ALB. Predictors of pressure ulcer risk in adult intensive care patients: A retrospective case-control study. Intensive Crit Care Nurs. 2018 Apr;45:6-10. doi: 10.1016/j.iccn.2017.09.007. Epub 2017 Dec 7. PMID 29223413
- [Background] Asghar M, Naseem S. Risk factors of pressure ulcer in elderly non-operative femur fracture patients. International Journal of Recent Scientific Research. 2018;9(7):28088-90.
- [Background] Kumar A, Sinha V. Comparative study of EUSOL and Silverstream in healing of pressure sore in traumatic spinal cord injury patients. International Journal of Orthopaedics. 2018;4(1):228-34.
- See also: Palese, Alvisa, et al. "What is the healing time of stage II pressure ulcers? findings from a secondary analysis." Advances in skin & wound care 28.2 (2015): 69-75. — https://journals.lww.com/aswcjournal/abstract/2015/02000/what_is_the_healing_time_of_stage_ii_pressure.5.aspx
- See also: Al-Hashemi, H., Alqurashi, K., Jan, R., Farran, A., Al-Sabban, B., & Thomson, J. (2019). Incidence, prevalence, and complications of pressure ulcers in general medical and surgical units using a multidisciplinary model (Prospective cohort). Biomedical Jo — https://ideas.repec.org/a/abf/journl/v18y2019i1p13340-13343.html
- See also: Haesler E, editor. National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel and Pan Pacific Pressure Injury Alliance. Prevention and Treatment of Pressure Ulcers: Quick Reference Guide. Osborne Park, Australia: Cambridge Media; 2014 — https://psmf.org/protected-content/
- See also: Related Info — https://www.nzwcs.org.nz/images/International_PUG/Quick_Reference_Guide_DIGITAL-PPPIA-Jan2016.pdf

DOCUMENTS (2):
  • Study Protocol (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT07193849/Prot_000.pdf
  • Informed Consent Form (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT07193849/ICF_001.pdf